CLINICAL TRIAL: NCT01955889
Title: Mobile Health Technology to Promote Physical Activity in Persons With Parkinson Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston University Charles River Campus (Other)
Responsible Party: Principal Investigator, Theresa D Ellis, Assistant Professor and Director of Center for Neurorehabilitation, Boston University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: BU-SAR-635
Record Dates: First submitted 2013-09-24; First posted 2013-10-08 (Estimated); Last update posted 2017-07-19 (Actual); Status verified 2017-07

CONDITIONS: Parkinson Disease
Keywords: Exercise; Rehabilitation; Telemedicine
MeSH Terms: conditions — Parkinson Disease; Motor Activity | interventions — Walking

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Mobile Health Technology (Experimental): Stretching and strengthening exercises provided via video using mobile health technology; walk daily using a pedometer; interact with a physical therapist remotely through an exercise application on a tablet device over 12 month period
  Interventions: Behavioral: Mobile Health Technology; Behavioral: Stretching & Strengthening Exercises; Behavioral: Walking with Pedometer
- Control (Active Comparator): Stretching and strengthening exercises provided using printed photographs; walk daily using a pedometer; interact with a physical therapist at the beginning of the 12 month study; no use of mobile technology
  Interventions: Behavioral: Stretching & Strengthening Exercises; Behavioral: Walking with Pedometer

INTERVENTIONS:
Behavioral: Mobile Health Technology
  Arms: Mobile Health Technology
Behavioral: Stretching & Strengthening Exercises
Behavioral: Walking with Pedometer

SUMMARY:
Persons with Parkinson Disease (PD) face significant declines in function resulting in greater disability. Function can improve through participation in exercise, yet many people with PD are physically inactive. Given that people with PD live long lifespans following diagnosis; it is essential to include routine exercise into their lives over the long-term. Physical therapy is effective in improving function in persons with PD. However, participation in on-going physical therapy indefinitely is not a realistic option due to limited healthcare resources. Interventions using mobile health technologies allow physical therapists to stay connected to patients over time potentially improving their ability to meet the changing needs of patients with PD. Innovative approaches using mobile health technology may improve outcome; however, the effectiveness of different approaches to improve function and reduce disability in PD is unknown.

The purpose of this study is to compare the effectiveness of two interventions to improve function and health-related quality of life in 65 people with PD. In one study group, participants receive a home exercise program, in written format, to continue on an independent basis. In the other study group, participants are instructed to continue with an exercise program, in their home, delivered using videos of the exercises on a computer tablet device. This use of mobile-Health technology allows the physical therapist to remotely monitor participants' progress and modify the exercise program to meet the changing needs of each patient. The long-term objective of this research is to determine the most efficient and effective way to improve function that can be widely disseminated to persons with PD.

ELIGIBILITY:
Inclusion Criteria:

* Inactive over the last 3 months
* Clinical diagnosis of idiopathic Parkinson's disease
* Mild to moderate disease severity
* Sufficient cognitive ability to follow study instructions
* Stable dose of Parkinson's medications for at least 2 weeks prior to study onset and during the 12 month study period unless medically necessary
* Able to walk without physical assistance or an assistive device for at least 6 continuous minutes
* Be interested in participating and provide informed consent

Exclusion Criteria:

* A diagnosis of atypical Parkinsonism
* Balance impairment (More than 2 falls in the previous month)
* Significant freezing
* Serious co-morbidities or medical conditions that may interfere with ability to participate in an exercise program (i.e., musculoskeletal, cardiovascular, and neurological (other than Parkinson's))

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2013-10; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in Physical Activity Level | 52-54 weeks
  Physical activity level will be assessed using an activity monitor worn around the ankle over a 7-day period at the beginning and the end of the study

SECONDARY OUTCOMES:
Change from Baseline in BriefBEST Balance Test | 52-54 weeks
  The BriefBEST balance test assesses balance using a series of tasks such as sitting and leaning, standing on compliant and non-compliant surfaces, stepping to the side, and walking on level surfaces
Change from Baseline in Six Minute Walk Test | 52-54 weeks
  Six Minute Walk Test is measure of the distance a participant is able to walk in a 6 minute time period
Change from Baseline in Falls Self-Efficacy Scale International | 52-54 weeks
  Falls Self-Efficacy Scale International is a self-administered questionnaire to assess the level of confidence in performing a series of 16 daily activities without falling
Change from Baseline in Unified Parkinson's Disease Rating Scale | 52-54 weeks
  Unified Parkinson's Disease Rating Scale assesses disability level related to the non-motor and motor signs in people with Parkinson's disease.
Change from Baseline in Parkinson's Disease Questionnaire-39 | 52-54 weeks
  Parkinson's Disease Questionnaire-39 is a self-administered questionnaire to assess the quality of life in people with Parkinson's disease
Change from Baseline in Self-Efficacy Exercise Scale | 52-54 weeks
  Self-Efficacy Exercise Scale is a self-administered questionnaire to assess confidence in ability to exercise
Change from Baseline in Functional Gait Assessment | 52-54 weeks
  Functional Gait Assessment assesses balance using a series of walking tasks, including walking in different directions, speeds, and around obstacles, including navigating stairs
Change from Baseline in Fatigue Severity Scale | 52-54 weeks
  Fatigue Severity Scale is a self-administered questionnaire where subjects are instructed to rate the impact of fatigue in their daily life over the prior week
Change from Baseline in Geriatric Depression Scale | 52-54 weeks
  Geriatric Depression Scale is a self-administered questionnaire to assess depression in individuals
Change from Baseline Apathy Scale | 52-54 weeks
  Apathy Scale is a self-administered questionnaire to assess apathy
Change from Baseline in Godin Leisure-Time Exercise Questionnaire | 52-54 weeks
  Godin Leisure-Time Exercise Questionnaire a self-administered questionnaire about the subjects leisure-time exercise habits over a typical seven day period

CONTACTS AND LOCATIONS:
Overall Officials: Terry Ellis, PhD, PT, NCS, Principal Investigator — Boston University; Nancy Latham, PhD, PT, Principal Investigator — Boston University
Locations (1):
- Center for Neurorehabilitation, College of Health & Rehabilitation Sciences, Sargent College, Boston University, Boston, Massachusetts, United States

REFERENCES:
- [Background] Kohl HW 3rd, Craig CL, Lambert EV, Inoue S, Alkandari JR, Leetongin G, Kahlmeier S; Lancet Physical Activity Series Working Group. The pandemic of physical inactivity: global action for public health. Lancet. 2012 Jul 21;380(9838):294-305. doi: 10.1016/S0140-6736(12)60898-8. PMID 22818941
- [Background] Shulman LM, Gruber-Baldini AL, Anderson KE, Vaughan CG, Reich SG, Fishman PS, Weiner WJ. The evolution of disability in Parkinson disease. Mov Disord. 2008 Apr 30;23(6):790-6. doi: 10.1002/mds.21879. PMID 18361474
- [Background] Rimmer JH, Marques AC. Physical activity for people with disabilities. Lancet. 2012 Jul 21;380(9838):193-5. doi: 10.1016/S0140-6736(12)61028-9. No abstract available. PMID 22818934
- [Background] Speelman AD, van de Warrenburg BP, van Nimwegen M, Petzinger GM, Munneke M, Bloem BR. How might physical activity benefit patients with Parkinson disease? Nat Rev Neurol. 2011 Jul 12;7(9):528-34. doi: 10.1038/nrneurol.2011.107. PMID 21750523
- [Background] Sisson SB, Camhi SM, Tudor-Locke C, Johnson WD, Katzmarzyk PT. Characteristics of step-defined physical activity categories in U.S. adults. Am J Health Promot. 2012 Jan-Feb;26(3):152-9. doi: 10.4278/ajhp.100326-QUAN-95. PMID 22208412
- [Background] Cavanaugh JT, Ellis TD, Earhart GM, Ford MP, Foreman KB, Dibble LE. Capturing ambulatory activity decline in Parkinson's disease. J Neurol Phys Ther. 2012 Jun;36(2):51-7. doi: 10.1097/NPT.0b013e318254ba7a. PMID 22592060
- [Background] Tomlinson CL, Patel S, Meek C, Clarke CE, Stowe R, Shah L, Sackley CM, Deane KH, Herd CP, Wheatley K, Ives N. Physiotherapy versus placebo or no intervention in Parkinson's disease. Cochrane Database Syst Rev. 2012 Aug 15;(8):CD002817. doi: 10.1002/14651858.CD002817.pub3. PMID 22895932
- [Background] Ellis T, Cavanaugh JT, Earhart GM, Ford MP, Foreman KB, Fredman L, Boudreau JK, Dibble LE. Factors associated with exercise behavior in people with Parkinson disease. Phys Ther. 2011 Dec;91(12):1838-48. doi: 10.2522/ptj.20100390. Epub 2011 Oct 14. PMID 22003171
- [Background] Ellis T, Boudreau JK, DeAngelis TR, Brown LE, Cavanaugh JT, Earhart GM, Ford MP, Foreman KB, Dibble LE. Barriers to exercise in people with Parkinson disease. Phys Ther. 2013 May;93(5):628-36. doi: 10.2522/ptj.20120279. Epub 2013 Jan 3. PMID 23288910
- [Background] Ellis T, Latham NK, DeAngelis TR, Thomas CA, Saint-Hilaire M, Bickmore TW. Feasibility of a virtual exercise coach to promote walking in community-dwelling persons with Parkinson disease. Am J Phys Med Rehabil. 2013 Jun;92(6):472-81; quiz 482-5. doi: 10.1097/PHM.0b013e31828cd466. PMID 23552335
- [Background] Tudor-Locke C, Bassett DR Jr. How many steps/day are enough? Preliminary pedometer indices for public health. Sports Med. 2004;34(1):1-8. doi: 10.2165/00007256-200434010-00001. PMID 14715035
- [Background] Ellis T, de Goede CJ, Feldman RG, Wolters EC, Kwakkel G, Wagenaar RC. Efficacy of a physical therapy program in patients with Parkinson's disease: a randomized controlled trial. Arch Phys Med Rehabil. 2005 Apr;86(4):626-32. doi: 10.1016/j.apmr.2004.08.008. PMID 15827910
- [Background] Watson A, Bickmore T, Cange A, Kulshreshtha A, Kvedar J. An internet-based virtual coach to promote physical activity adherence in overweight adults: randomized controlled trial. J Med Internet Res. 2012 Jan 26;14(1):e1. doi: 10.2196/jmir.1629. PMID 22281837
- [Background] Ellis T, Cavanaugh JT, Earhart GM, Ford MP, Foreman KB, Dibble LE. Which measures of physical function and motor impairment best predict quality of life in Parkinson's disease? Parkinsonism Relat Disord. 2011 Nov;17(9):693-7. doi: 10.1016/j.parkreldis.2011.07.004. Epub 2011 Aug 5. PMID 21820940
- [Background] Muslimovic D, Post B, Speelman JD, Schmand B, de Haan RJ; CARPA Study Group. Determinants of disability and quality of life in mild to moderate Parkinson disease. Neurology. 2008 Jun 3;70(23):2241-7. doi: 10.1212/01.wnl.0000313835.33830.80. PMID 18519873
- [Background] Shulman LM. Understanding disability in Parkinson's disease. Mov Disord. 2010;25 Suppl 1:S131-5. doi: 10.1002/mds.22789. PMID 20187231
- [Background] Resnick B, Nahm ES, Orwig D, Zimmerman SS, Magaziner J. Measurement of activity in older adults: reliability and validity of the Step Activity Monitor. J Nurs Meas. 2001 Winter;9(3):275-90. PMID 11881269
- [Background] Schmidt AL, Pennypacker ML, Thrush AH, Leiper CI, Craik RL. Validity of the StepWatch Step Activity Monitor: preliminary findings for use in persons with Parkinson disease and multiple sclerosis. J Geriatr Phys Ther. 2011 Jan-Mar;34(1):41-5. doi: 10.1519/JPT.0b013e31820aa921. PMID 21937891
- [Background] Speelman AD, van Nimwegen M, Borm GF, Bloem BR, Munneke M. Monitoring of walking in Parkinson's disease: validation of an ambulatory activity monitor. Parkinsonism Relat Disord. 2011 Jun;17(5):402-4. doi: 10.1016/j.parkreldis.2011.02.006. Epub 2011 Mar 1. No abstract available. PMID 21367643
- [Background] Tickle-Degnen L, Ellis T, Saint-Hilaire MH, Thomas CA, Wagenaar RC. Self-management rehabilitation and health-related quality of life in Parkinson's disease: a randomized controlled trial. Mov Disord. 2010 Jan 30;25(2):194-204. doi: 10.1002/mds.22940. PMID 20077478
- [Derived] Ellis TD, Cavanaugh JT, DeAngelis T, Hendron K, Thomas CA, Saint-Hilaire M, Pencina K, Latham NK. Comparative Effectiveness of mHealth-Supported Exercise Compared With Exercise Alone for People With Parkinson Disease: Randomized Controlled Pilot Study. Phys Ther. 2019 Feb 1;99(2):203-216. doi: 10.1093/ptj/pzy131. PMID 30715489
- See also: Center for Neurorehabilitation at Boston University — http://www.bu.edu/neurorehab/research/